CLINICAL TRIAL: NCT01637610
Title: Detection of Preterm Prelabour Rupture of Membranes With AmniSure Placental Alpha Macroglobulin-1 Rapid Immunoassay
Brief Title: Detection of PPROM With AmniSure PAMG-1 Rapid Immunoassay
Status: Terminated | Type: Observational
Why Stopped: Lack of support with enrollment.
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Sabrina Stewart, Principal Investigator, University of Saskatchewan
Other Study IDs: 11-67
Record Dates: First submitted 2012-06-28; First posted 2012-07-11 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2012-07

CONDITIONS: Preterm Premature Rupture of Fetal Membranes
Keywords: placental alpha microglobulin-1; AmniSure; preterm; rupture of fetal membranes
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PPROM: All women presenting to assessment at the labour and delivery unit at RUH with suspected PPROM between 16+0 and 36+6 weeks gestation.

SUMMARY:
The investigators will test the hypothesis that in a preterm population with a gestational age of 16+0 and 36+6 weeks AmniSure PAMG-1 rapid immunoassay will be more accurate than conventional methods (speculum examination for combination of pooling, nitrazine and ferning) for the detection of Preterm Prelabour Rupture of Membranes (PROM).

DETAILED DESCRIPTION:
Prior studies of AmniSure have included a heterogeneous population of women with preterm and term pregnancies.10-12 No study to date has specifically addressed and been powered to detect the efficacy of AmniSure in pregnancies between 16+0 and 36+6 weeks. The objective of the proposed research is to evaluate the usefulness of AmniSure PAMG-1 rapid immunoassay in the evaluation of preterm prelabour rupture of membranes (PPROM) compared to standard detection of PPROM with a speculum examination for combination of pooling, nitrazine and ferning.

ELIGIBILITY:
Inclusion Criteria:

* women presenting to assessment at the labour and delivery unit at RUH with suspected PPROM between 16+0 and 36+6 weeks gestation
* consent to enrollment

Exclusion Criteria:

* vaginal bleeding
* active labor (cervical dilation > 2 cm or effacement > 80%)
* multiple pregnancy
* fetal anomalies
* placenta previa
* fluid loss per vagina > 7 days
* prior inclusion in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women presenting to assessment at the labour and delivery unit at RUH with suspected PPROM between 16+0 and 36+6 weeks gestation.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
accuracy of Amnisure vs conventional testing for PPROM | up to 24 weeks
  After delivery, the charts will be reviewed and information will be used to determine the final diagnosis of membrane status as ruptured or intact on initial presentation and will be used to evaluate the accuracy of the AmniSure test results.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal University Hopsital, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Lee SM, Romero R, Park JW, Kim SM, Park CW, Korzeniewski SJ, Chaiworapongsa T, Yoon BH. The clinical significance of a positive Amnisure test in women with preterm labor and intact membranes. J Matern Fetal Neonatal Med. 2012 Sep;25(9):1690-8. doi: 10.3109/14767058.2012.657279. Epub 2012 Apr 25. PMID 22280400
- [Background] Abdelazim IA, Makhlouf HH. Placental alpha microglobulin-1 (AmniSure((R)) test) for detection of premature rupture of fetal membranes. Arch Gynecol Obstet. 2012 Apr;285(4):985-9. doi: 10.1007/s00404-011-2106-4. Epub 2011 Oct 30. PMID 22037683
- [Background] Lee SM, Lee J, Seong HS, Lee SE, Park JS, Romero R, Yoon BH. The clinical significance of a positive Amnisure test in women with term labor with intact membranes. J Matern Fetal Neonatal Med. 2009 Apr;22(4):305-10. doi: 10.1080/14767050902801694. PMID 19350444
- [Background] Cousins LM, Smok DP, Lovett SM, Poeltler DM. AmniSure placental alpha microglobulin-1 rapid immunoassay versus standard diagnostic methods for detection of rupture of membranes. Am J Perinatol. 2005 Aug;22(6):317-20. doi: 10.1055/s-2005-870896. PMID 16118720